CLINICAL TRIAL: NCT01347528
Title: A Randomized, Controlled Trial Using a TELEmedicine Solution to Improve MEDication Adherence in Chronic Heart Failure (TELEMED-HF)
Brief Title: Improving MEDication Adherence in Chronic Heart Failure Using a TELEmedicine Device (TELEMED-HF)
Acronym: TELEMED-HF
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: logistic and financial accounting reasons
Sponsor: Tilburg University (Other)
Collaborators: The Elisabeth-TweeSteden Hospital (Other)
Responsible Party: Principal Investigator, Nina Kupper PhD, Nina Kupper, PhD, Tilburg University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UVT MP 002
Record Dates: First submitted 2011-04-29; First posted 2011-05-04 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Heart Failure
Keywords: Medication adherence; Heart failure; Telemonitoring; Determinants of adherence
MeSH Terms: conditions — Heart Failure; Medication Adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TELEmonitoring intervention (Experimental)
  Interventions: Behavioral: Medication Adherence Support System (MASS)
- Usual care (No Intervention)

INTERVENTIONS:
Behavioral: Medication Adherence Support System (MASS) — The intervention consists of the use of an electronic Medication Adherence Monitor for a 6-month period as well as 2 visits to the heart failure outpatient clinic of the TweeSteden hospital (usual care). This monitor (a) dispenses all prescribed medication in the right dosage at the specified time, (b) reminds patients to take their medications through an alarm, sms or voicemail service and records adherence, and (c) sends critical data about non-adherence to the heart failure nurse, via a web application (CarebyWeb). The Medication Adherence Monitor is provided to the patient by the hospital pharmacy, including an instruction how to use the device. After the intervention patients return to usual care only. We expect a training effect, with continued improved adherence in the intervention group.
  Other Names: PICO® by Vitaphone Nederland BV
  Arms: TELEmonitoring intervention

SUMMARY:
TELEMED-HF is a randomized, controlled clinical intervention trial designed to: (1) examine the efficacy of an electronic Medication Adherence Support System (MASS) in improving and monitoring patients' medication adherence; to (2) i determine the effect of medication adherence on hospitalization and health care consumption.

ELIGIBILITY:
Inclusion Criteria:

* Stable systolic heart failure
* New York Heart Association functional class II-III, with a decreased pump function (left ventricular ejection fraction (LVEF) <45%)
* Titrated to the most optimal doses of ACE-inhibitor or Angiotensin Receptor Blocker, and beta-blocker
* Receiving stable doses of at least 3 heart failure medications (at multiple times during the day) for 1 month with no plans to add or adjust heart failure medications or titrate further in the immediate future.

Exclusion Criteria:

* Age younger than 50 years
* Diastolic heart failure (intact pump function)
* Myocardial infarction, invasive treatment (percutaneous coronary intervention (PCI) or coronary artery bypass grafting (CABG)), or hospitalization within 1 month prior to inclusion
* Life-threatening comorbid conditions (e.g., cancer)
* Diminished mental capacities (suspected cognitive decline will be confirmed by a mini mental state examination (MMSE))
* History of psychiatric disorders apart from affective disorders (depression and anxiety disorders)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-10; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Change in medication adherence | Baseline, 6 months, 9 months, 12 months, 15 months, and 18 months
  Objective medication adherence will be assessed using the MASS monitor output collected in a web-based application and the refill rates provided by the patients' pharmacies.
Change in number of hospitalizations (costs) | Baseline, 6 months, 9 months, 12 months, 15 months, and 18 months
  A cost-benefit analysis will be assessed by means of the TiC-P questionnaire and event rate (and related DBC (diagnosis treatment combination, the Dutch system to allocate costs to treatments of specific patient groups)). The TiC-P questionnaire will enable us to compare healthcare consumption in the intervention and control group.

SECONDARY OUTCOMES:
Change in self-care behavior and Quality of Life | Baseline, 6 months, 12 months, and 18 months
Course of disease severity | Baseline, 6 months, 12 months, and 18 months
  Clinical characteristics (e.g. NYHA function class determination, LVEF, exercise capacity, blood tests) and self-reported HF symptoms
Change in psychological variables | Baseline, 6 months, 12 months, and 18 months
  Type D personality, depression, anxiety

CONTACTS AND LOCATIONS:
Overall Officials: Nina Kupper, Principal Investigator — Tilburg University, The Netherlands
Locations (1):
- TweeSteden Hospital, Tilburg, North Brabant, Netherlands

REFERENCES:
- [Derived] Kessing D, Denollet J, Widdershoven J, Kupper N. Investigating a TELEmedicine solution to improve MEDication adherence in chronic Heart Failure (TELEMED-HF): study protocol for a randomized controlled trial. Trials. 2011 Oct 14;12:227. doi: 10.1186/1745-6215-12-227. PMID 21999637